CLINICAL TRIAL: NCT00001304
Title: Treatment of Hypoparathyroidism With Synthetic Human Parathyroid Hormone 1-34
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Karen K. Winer, M.D., medical officer, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 920011; 92-CH-0011 (Other Grant/Funding Number: NIH Clinical Center_NICHD)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; Parathyroid Hormone; Vitamin D; Calcium Metabolism; PTH 1-34; Bone
MeSH Terms: conditions — Hypoparathyroidism | interventions — Calcitriol; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTH 1-34 (Experimental): All patients received twice daily synthetic Human Parathyroid Hormone 1-34.
  Interventions: Drug: Synthetic Human Parathyroid Hormone 1-34
- Calcitriol & Calcium (Experimental): All patients received twice daily Calcitriol and Calcium 1000mg divided into four doses daily.
  Interventions: Drug: Calcitriol & Calcium

INTERVENTIONS:
Drug: Synthetic Human Parathyroid Hormone 1-34 — twice daily subcutaneous injections
  Other Names: teriperitide
  Arms: PTH 1-34
Drug: Calcitriol & Calcium — Twice daily oral calcitriol with 1000 mg Calcium carbonate supplementation
  Other Names: rocaltrol; 1,25 OH Vitamin D
  Arms: Calcitriol & Calcium

SUMMARY:
This study has been important in establishing synthetic human parathyroid hormone 1-34 (PTH) as a beneficial treatment for hypoparathyroidism, superior to conventional therapy with calcium and calcitriol. Providing synthetic human parathyroid hormone 1-34 (PTH) to patients who are unresponsive to conventional therapy has enabled severe cases of hypoparathyroidism to be managed effectively with the investigational drug, PTH. The primary goals of this study are to (1) provide long-term PTH therapy to patients who do not respond to conventional therapy; (2) understand the long-term effect of therapeutic PTH replacement on kidney function and bone mineral density; (3) study and track linear growth and bone accrual in children with hypoparathyroidism. (4) determine if subjects reach a normal level of peak bone mass and if the timing of this is comparable to normal age-matched healthy controls.

DETAILED DESCRIPTION:
Vitamin D and its analogs, the conventional treatment for hypoparathyroidism, are associated with chronic hypercalciuria due to their lack of calcium-retaining effect in the kidney. This side effect usually occurs even while maintaining the serum calcium in the normal range and may lead to calcium deposition in the kidney (nephrocalcinosis) and renal insufficiency. This study examines the long-term effects of subcutaneous parathyroid hormone (PTH) therapy on calcium metabolism, bone, and renal function. Our previous short-term pilot study comparing subcutaneous PTH with calcitriol demonstrated a significant decrease in urinary calcium excretion during PTH therapy. Based upon these results, we hypothesized that treatment with PTH is more physiologic and provides improved long-term metabolic control. Additionally, treatment with PTH may avoid the adverse side effects on the kidney that are associated with conventional therapy. Patients initially come to the Clinical Center for a two week inpatient evaluation. Subsequent follow-up will occur semiannually on an outpatient basis.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will include patients (ages 17-69) with biochemically confirmed hypoparathyroidism.

EXCLUSION CRITERIA

Women who are pregnant will be excluded.

Ages: 17 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1991-10; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Winer, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Winer KK, Yanovski JA, Cutler GB Jr. Synthetic human parathyroid hormone 1-34 vs calcitriol and calcium in the treatment of hypoparathyroidism. JAMA. 1996 Aug 28;276(8):631-6. PMID 8773636
- [Background] Winer KK, Yanovski JA, Sarani B, Cutler GB Jr. A randomized, cross-over trial of once-daily versus twice-daily parathyroid hormone 1-34 in treatment of hypoparathyroidism. J Clin Endocrinol Metab. 1998 Oct;83(10):3480-6. doi: 10.1210/jcem.83.10.5185. PMID 9768650
- [Background] Winer KK, Zhang B, Shrader JA, Peterson D, Smith M, Albert PS, Cutler GB Jr. Synthetic human parathyroid hormone 1-34 replacement therapy: a randomized crossover trial comparing pump versus injections in the treatment of chronic hypoparathyroidism. J Clin Endocrinol Metab. 2012 Feb;97(2):391-9. doi: 10.1210/jc.2011-1908. Epub 2011 Nov 16. PMID 22090268
- [Background] Winer KK, Ko CW, Reynolds JC, Dowdy K, Keil M, Peterson D, Gerber LH, McGarvey C, Cutler GB Jr. Long-term treatment of hypoparathyroidism: a randomized controlled study comparing parathyroid hormone-(1-34) versus calcitriol and calcium. J Clin Endocrinol Metab. 2003 Sep;88(9):4214-20. doi: 10.1210/jc.2002-021736. PMID 12970289
- [Background] Winer KK, Sinaii N, Peterson D, Sainz B Jr, Cutler GB Jr. Effects of once versus twice-daily parathyroid hormone 1-34 therapy in children with hypoparathyroidism. J Clin Endocrinol Metab. 2008 Sep;93(9):3389-95. doi: 10.1210/jc.2007-2552. Epub 2008 May 20. PMID 18492754

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcitriol and Calcium: Twice daily po calcitriol with calcium carbonate given 4 times daily
- PTH 1-34: PTH 1-34 given as 2 subcutaneous injections daily
Period: Overall Study
Arm/Group | Calcitriol and Calcium | PTH 1-34
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcitriol and Calcium | PTH 1-34 | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Serum 1,25-hydroxyvitamin D Level
Description: Measurements were taken 1 hour before the morning dose of PTH or, calcitriol and calcium; UOM = pg/ml. Measurements were obtained on three successive days (three separate measures) semiannually at the NIH CC for each protocol subject. The average data are the average of these three semi-annual data points for each subject which are then averaged across all the semi-annual means for all subjects within each arm over the three years of study.
Time Frame: 3 years
Population: All patients on the study
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Calcitriol and Calcium | PTH 1-34
Number analyzed (Participants) | 13 | 14
pg/ml | 40 (5) | 43 (5)

2. Secondary Outcome: Serum 25-hydroxyvitamin D Level
Description: Measurements were taken 1 hour before the morning dose of PTH or, calcitriol and calcium; UOM = ng/ml. Measurements were obtained on three successive days (three separate measures) semiannually at the NIH CC for each protocol subject. The average data are the average of these three semi-annual data points for each subject which are then averaged across all the semi-annual means for all subjects within each arm over the three years of study.
Time Frame: 3 years
Population: All patients on the study
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Calcitriol and Calcium | PTH 1-34
Number analyzed (Participants) | 13 | 14
ng/ml | 31 (5) | 28 (4)

3. Primary Outcome: Serum Calcium Level
Description: Measurements were taken 1 hour before the morning dose of PTH or, calcitriol and calcium; UOM = mmol/liter, normal range 2.05-2.5. Measurements were obtained on three successive days (three separate measures) semiannually at the NIH CC for each protocol subject. The average data are the average of these three semi-annual data points for each subject which are then averaged across all the semi-annual means for all subjects within each arm over the three years of study.
Time Frame: 3 years
Population: All patients on the study
Measure: Mean (Standard Deviation); unit: mmol/liter
Arm/Group | Calcitriol and Calcium | PTH 1-34
Number analyzed (Participants) | 13 | 14
mmol/liter | 2 (0.01) | 1.92 (0.02)

4. Secondary Outcome: Serum Magnesium Level
Description: Measurements were taken 1 hour before the morning dose of PTH or, calcitriol and calcium; UOM = mmol/liter, normal range 0.65-1.05. Measurements were obtained on three successive days (three separate measures) semiannually at the NIH CC for each protocol subject. The average data are the average of these three semi-annual data points for each subject which are then averaged across all the semi-annual means for all subjects within each arm over the three years of study.
Time Frame: 3 years
Population: All patients on the study
Measure: Mean (Standard Deviation); unit: mmol/liter
Arm/Group | Calcitriol and Calcium | PTH 1-34
Number analyzed (Participants) | 13 | 14
mmol/liter | 0.75 (0.01) | 0.73 (0.02)

5. Secondary Outcome: Serum Phosphorus Level
Description: Measurements were taken 1 hour before the morning dose of PTH or, calcitriol and calcium; UOM = mmol/liter, normal range 0.7-1.4. Measurements were obtained on three successive days (three separate measures) semiannually at the NIH CC for each protocol subject. The average data are the average of these three semi-annual data points for each subject which are then averaged across all the semi-annual means for all subjects within each arm over the three years of study.
Time Frame: 3 years
Population: All patients on the study
Measure: Mean (Standard Deviation); unit: mmol/liter
Arm/Group | Calcitriol and Calcium | PTH 1-34
Number analyzed (Participants) | 13 | 14
mmol/liter | 4.5 (0.05) | 4.6 (0.08)

6. Secondary Outcome: Urinary Creatinine Clearance
Description: Measurements were taken 1 hour before the morning dose of PTH or, calcitriol and calcium; UOM = ml/min, normal range 90-125. Measurements were obtained on three successive days (three separate measures) semiannually at the NIH CC for each protocol subject. The average data are the average of these three semi-annual data points for each subject which are then averaged across all the semi-annual means for all subjects within each arm over the three years of study.
Time Frame: 3 years
Population: All patients on the study
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Calcitriol and Calcium | PTH 1-34
Number analyzed (Participants) | 13 | 14
ml/min | 84 (13) | 80 (10)

7. Primary Outcome: Urine Calcium Excretion Level
Description: Measurements were taken1 hour before the morning dose of PTH or, calcitriol and calcium; UOM = mmol/24 h, normal range 1.25-6.25. Measurements were obtained on three successive days (three separate measures) semiannually at the NIH CC for each protocol subject. The average data are the average of these three semi-annual data points for each subject which are then averaged across all the semi-annual means for all subjects within each arm over the three years of study.
Time Frame: 3 years
Population: All patients on the study
Measure: Mean (Standard Deviation); unit: mmol/24 h
Arm/Group | Calcitriol and Calcium | PTH 1-34
Number analyzed (Participants) | 13 | 14
mmol/24 h | 8.2 (0.51) | 5.8 (0.27)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- PTH 1-34: All patients received twice daily synthetic Human Parathyroid Hormone 1-34.
  PTH 1-34
- Calcitriol & Calcium: All patients received twice daily Calcitriol and Calcium 1000mg divided into four doses daily.
  Calcitriol & Calcium
Arm/Group | PTH 1-34 | Calcitriol & Calcium
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

LIMITATIONS AND CAVEATS:
Study reported here was the primary long-term study for adults with hypoparathyroidism. Subsequent studies included additional patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes